CLINICAL TRIAL: NCT02350998
Title: A 1-Month, Prospective, Multicenter, Open-Label Study of OTO-201 Given as a Single Trans-Tympanic Tube Administration for Intra-Operative Treatment of Middle Ear Effusion in Pediatric Subjects With Otitis Media Requiring Tympanostomy Tube Placement
Brief Title: Open-Label Study of OTO-201 for Middle Ear Effusion Evaluating Trans-Tympanostomy Tube Administration
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otonomy, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201-201404
Record Dates: First submitted 2015-01-21; First posted 2015-01-30 (Estimated); Results first posted 2020-09-23 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Bilateral Middle Ear Effusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OTO-201 (Experimental): 6 mg OTO-201 administered trans-tympanostomy tube
  Interventions: Drug: OTO-201

INTERVENTIONS:
Drug: OTO-201

SUMMARY:
This is a 1-month, prospective, multicenter, open-label study in pediatric subjects with bilateral middle ear effusion requiring tympanostomy tube placement. Eligible subjects will receive a single dose to each ear of 6 mg OTO-201, administered intraoperatively into the middle ear through the lumen of the tympanostomy tube (trans-tympanostomy tube TTT). The study is designed to characterize safety and any procedural issues associated with TTT drug administration of OTO-201.

ELIGIBILITY:
Inclusion Criteria includes, but is not limited to:

* Subject is a male or female aged 6 months to 17 years, inclusive
* Subject has a clinical diagnosis of bilateral middle ear effusion requiring tympanostomy tube placement
* Subject's caregiver is willing to comply with the protocol an attend all study visits

Exclusion Criteria includes, but is not limited to:

* Subject has a history of prior ear or mastoid surgery, not including myringotomy or myringotomy with tympanostomy tube placement
* Subject has a history of sensorineural hearing loss
* Subject has been designated for any other surgical procedure that would occur concurrently with TT placement, such as, but not limited to adenoidectomy or tonsillectomy

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2015-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl LeBel, PhD, Study Chair — Otonomy, Inc.
Locations (5):
- United States (5):
  - Central California Ear, Nose and Throat, Fresno, California
  - Charlotte Eye, Ear, Nose and Throat Associates, Charlotte, North Carolina
  - Charlotte Eye, Ear, Nose and Throat Associates, Matthews, North Carolina
  - Piedmont Ear, Nose and Throat, Winston-Salem, North Carolina
  - Carolina Ear, Nose and Throat, Orangeburg, South Carolina

RESULTS

PARTICIPANT FLOW:
Groups:
- 6 mg OTO-201: 6 mg ciprofloxacin: single Trans-Tympanic Tube Administration
Period: Overall Study
Arm/Group | 6 mg OTO-201
Started | 33
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 6 mg OTO-201
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 33
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.92 (2.465)
Age, Customized [Count of Participants; unit: Participants]
  6 months to 2 years | 17
  >2 years | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 23
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Otoscopic Examination: Auricle and Meatus
Description: Number of ears whose external ear and ear canal (auricle and meatus), when examined through an otoscope, appeared normal at Baseline and appeared abnormal at Day 29
Time Frame: Up to 1 month
Population: Safety analysis set : consisted of all enrolled and treated subjects
Measure: Count of Units; unit: ears
Units Other Than Participants: ears
Groups:
- 6mg OTO-201: 6 mg ciprofloxacin: single Trans-Tympanic Tube Administration
Arm/Group | 6mg OTO-201
Number analyzed (Participants) | 33
Number analyzed (ears) | 66
ears | 1

2. Primary Outcome: Otoscopic Examination: Tympanic Membrane
Description: Number of ears whose ear drum (tympanic membrane), when examined through an otoscope, appeared normal at Baseline and appeared abnormal at Day 29
Time Frame: up to 1 month
Population: Safety analysis set: all enrolled and treated subjects
Measure: Count of Units; unit: ears
Units Other Than Participants: ears
Arm/Group | 6 mg OTO-201
Number analyzed (Participants) | 33
Number analyzed (ears) | 66
ears | 2

3. Primary Outcome: Otoscopic Examination: Tube Patency
Description: Subjects with at least one ear tube patent (i.e., not blocked) at Day 29
Time Frame: Up to 1 month
Population: Safety analysis set: all enrolled and treated subjects
Measure: Count of Participants; unit: Participants
Arm/Group | 6 mg OTO-201
Number analyzed (Participants) | 33
Participants | 32

4. Secondary Outcome: Feasibility of Administration
Description: Ease of administering OTO-201 through the tympanostomy tube: Number of subjects that investigators rated ease of administration as either "easy" or "very easy"
Time Frame: Day 1
Population: Safety analysis set consisted of all enrolled and treated subjects
Measure: Count of Participants; unit: Participants
Groups:
- 6 mg OTO-201: 6 mg ciprofloxacin: single Trans-Tympanic Tube Admin istration
Arm/Group | 6 mg OTO-201
Number analyzed (Participants) | 33
Participants | 29

ADVERSE EVENTS:
Time Frame: Adverse events were reported during dosing and up to 1 month following dosing.
Arm/Group | 6 mg OTO-201
All-Cause Mortality (participants affected / at risk) | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 20/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 6 mg OTO-201 (N=33)
Nasopharyngitis (Infections and infestations) | 7
Upper Respiratory Infection (Infections and infestations) | 3
Ear Pain (Ear and labyrinth disorders) | 4
Pyrexia (General disorders) | 4
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication subject to Sponsor consent.